CLINICAL TRIAL: NCT04140383
Title: Outcomes of Cataract Surgeries in Patients With Advanced Age
Brief Title: Cataract Surgery In Patients With Advanced Age
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Burçin Çakır, Principal investigator, Sakarya University
Other Study IDs: Sakarya Ophthalmology
Record Dates: First submitted 2019-10-13; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Cataract Senile
Keywords: geriatry; cataract surgery; advanced age
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1, patients aged 85 years and older: 75 eyes of 75 patients (39 female, 36 male) Mean age: 86,8 ± 1,8 years
  Interventions: Procedure: Cataract Surgery
- Group 2, patients aged 65 and 85 years: 77 eyes of 77 patients (34 female, 43 male) Mean age:73,3 ± 5,2 years
  Interventions: Procedure: Cataract Surgery

INTERVENTIONS:
Procedure: Cataract Surgery — Cataract surgery was performed by using phacoemulsification technique, routinely. But other techniques for instance extra or intracapsular cataract extraction (ECCE, ICCE) techniques were performed when needed. Phacoemulsification technique was performed by 2 experienced surgeon (G.A. and E.C.) under topical anesthesia, thorough limbal incision. Foldable single piece hydrophobic acrylic intraocular lens (IOL) was inserted in the bag. In the presence of complications related to anterior or posterior capsules, 3 pieces IOL was preferred. When ECCE technique was chosen, single piece polymethyl methacrylate IOL was inserted.

SUMMARY:
This study evaluates and compares clinical outcomes of < 85 and ≥ 85 year old patients who underwent cataract surgeries.

DETAILED DESCRIPTION:
The medical records of patients who were underwent cataract surgery between January 2014 and October 2017 were investigated retrospectively and patients 65 years and older were recruited. Two groups were made according to age: group1 composed of patients age range between 65 and 85 years and group 2 composed of patients 85 years and older. Gender, presence of diabetes mellitus (DM), hypertension (HT), drug use were noted.

The results of best corrected visual acuity (BCVA) converted to LogMar, intraocular pressure (IOP) before and 3 months after operation, biomicroscopic and fundus examinations were investigated.

Additional ocular diseases such as glaucoma, age related macular degeneration (AMD), pseudoexfoliation syndrome, retinopathies and maculopathies related to systemic diseases were noted. Pupil dilation properties were also noted as poor, mid or full pupil dilation.

Cataract surgery techniques such as phacoemulsification, extra- and intracapsular lens extractions, peroperative complications, intracameral drug use were investigated.

these aforementioned outcomes evaluated and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 years and older patients who underwent cataract surgery

Exclusion Criteria:

* patients aged below 65 years who underwent cataract surgery

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: patients aged 65 years and older who underwent cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | Before cataract surgery
  Best corrected visual acuity converted to LogMar
Best corrected visual acuity | three months after cataract surgery
  Best corrected visual acuity converted to LogMar

SECONDARY OUTCOMES:
presence of Diabetes Mellitus | Baseline (Before cataract surgery)
  number of participants who have diabetes mellitus
presence of essential hypertension | before cataract surgery
  number of participants who have essential hypertension
oral acetylsalicylic acid use | before cataract surgery
  number of participants who have a history of acetylsalicylic acid use
oral flomax use | before cataract surgery
  number of participants who have a history of oral flomax use
presence of age related macular degeneration | Baseline (Before cataract surgery)
  number of participants who have age related macular degeneration
presence of glaucoma | before cataract surgery
  number of participants who have glaucoma
presence of pseudoexfoliation | before cataract surgery
  number of participants who have pseudoexfoliation
presence of poor pupil dilation | During cataract surgery
  number of participants who have poor pupil dilation
presence of zonule deficiency | During cataract surgery
  number of participants who have zonule deficiency
Cataract types in patients who underwent cataract surgery | Baseline (Before cataract surgery)
  number of participants who have nuclear, posterior subcapsular, corticonuclear, mature, nigra, traumatic cataract
measurement of effective phacoemulsification time | During cataract surgery
  measurement of effective phacoemulsification time in participants who underwent cataract surgery
presence of posterior capsule rupture | During cataract surgery
  participants who had posterior capsule rupture during surgery
anterior vitrectomy | during surgery
  number of participants who needed anterior vitrectomy during cataract surgery
presence of aphakia | 3 months after cataract surgery
  number of participants who left aphakic after cataract surgery
intracameral adrenalin use | during surgery
  number of participants who needed intracameral adrenalin use

CONTACTS AND LOCATIONS:
Overall Officials: Burcin Cakir, MD, Principal Investigator — Sakarya University
Locations (1):
- Sakarya University Ophthalmology Department, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Syam PP, Eleftheriadis H, Casswell AG, Brittain GP, McLeod BK, Liu CS. Clinical outcome following cataract surgery in very elderly patients. Eye (Lond). 2004 Jan;18(1):59-62. doi: 10.1038/sj.eye.6700521. PMID 14707968
- See also: Sussex Eye Hospital, Brighton, United Kingdom — http://rdcu.be/bUabz
- Available data/document: Clinical Study Report — http://rdcu.be/bUabz